CLINICAL TRIAL: NCT06692452
Title: A Phase II Study of Tazemetostat in Combination With CHOP for Previously Untreated T Cell Lymphoma
Brief Title: Tazemetostat Plus CHOP in 1L T-cell Lymphoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Ipsen requested a temporary closure due to a safety concern.
Sponsor: Eric Jacobsen, MD (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor-Investigator, Eric Jacobsen, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-462
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Peripheral T Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Enteropathy-Associated T-Cell Lymphoma; Monomorphic Epitheliotropic Intestinal T-Cell Lymphoma
Keywords: Lymphoma; Peripheral T-cell Lymphoma; PTCL; Angioimmunoblastic T-cell Lymphoma; AITL; Enteropathy-Associated T-Cell Lymphoma; EATL; Monomorphic Epitheliotropic Intestinal T-Cell Lymphoma; MEITL
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Peripheral; Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma | interventions — tazemetostat; Doxorubicin; Vincristine; Prednisone; Prednisolone; Cyclophosphamide; Carmustine; Etoposide; etoposide phosphate; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tazemetostat + CHOP Therapy + Transplant Elected (Experimental): Enrolled participants will complete:
  * Baseline visit
  * Prephase Period: Days -14 through -1: Predetermined dose of Tazemetost 2x daily
  * Induction Period: Cycles 1 through 6 (21 day cycles):
    * Cycle 1 Day 1: tumor biopsy and CT scan
    * Day 1: Predetermined dose of Cyclophosphamide once, Doxorubicin once, and Vincristine once
    * Days 1 through 5: Predetermined dose of Prednisone 1x daily
    * Days 2 through 21: Predetermined dose of Tazemetost 2x daily
    * Prior to Cycle 4 Day 1: Pet-CT scan
  * Note, treatment will stop if participants do not respond to the drugs after the first 3 cycles
  * Bone marrow biopsy and Pet-CT scan at end of Cycle 6
  * Maintenance Period:
  * Day 0: autologous stem cell transplant with BiCNU, Etoposide, Cytarabine, and Melphalan (BEAM)
  * Day 100: PET-CT scan
  * Cycles 1 through 6 (28 day cycles):
    --Days 1 through 28: Predetermined dose of Tazemetost 2x daily
  * After Cycle 3: CT scan
  * Cycle 4 Day 1: CT scan
  * End of treatment visit
  * Follow up is for 4 years
  Interventions: Drug: Tazemetostat; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Cytoxan; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan
- Tazemetostat + CHOP Therapy + Transplant Not Elected (Experimental): Enrolled participants will complete:
  * Baseline visit
  * Prephase Period: Days -14 through -1: Predetermined dose of Tazemetost 2x daily
  * Induction Period: Cycles 1 through 6 (21 day cycles):
    * Cycle 1 Day 1: tumor biopsy and CT scan
    * Day 1: Predetermined dose of Cyclophosphamide once, Doxorubicin once, and Vincristine once
    * Days 1 through 5: Predetermined dose of Prednisone 1x daily
    * Days 2 through 21: Predetermined dose of Tazemetost 2x daily
    * Prior to Cycle 4 Day 1: Pet-CT scan
  * Note, treatment will stop if participants do not respond to the drugs after the first 3 cycles
  * Pet-CT scan at end of Cycle 6.
  * Maintenance Period:
  * Cycles 1 through 6 (28 day cycles):
    --Days 1 through 28: Predetermined dose of Tazemetost 2x daily.
  * After Cycle 3: CT scan
  * Cycle 4 Day 1: CT scan
  * End of treatment visit
  * Follow up is for 4 years
  Interventions: Drug: Tazemetostat; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Cytoxan

INTERVENTIONS:
Drug: Tazemetostat — EZH2 inhibitor, 200 mg tablet, taken orally per protocol.
  Other Names: Tazverik; [1,1'-Biphenyl]-3-carboxamide,N-[(1,2-dihydro- 4,6-dimethyl-2-oxo-3-pyridinyl)methyl]-5- [ethyl(tetrahydro-2H-pyran-4-yl)amino]-4-methyl- 4'-(4-morpholinylmethyl)-, hydrobromide (1:1)
Drug: Doxorubicin — Anthracycline antibiotic, 10, 20, 50, 100, and 200 mg vials, via intravenous (into the vein) infusion per institutional standard of care.
  Other Names: Hydroxydaunorubicin
Drug: Vincristine — Vinca Alkaloid, 1, 2, and 5mL vials, via intravenous (into the vein) infusion per institutional standard of care.
  Other Names: Oncovin
Drug: Prednisone — Corticosteroid, 1, 2.5, 5, 10, 20, 25, and 50 mg tablets, taken orally per institutional standard of care.
  Other Names: Prednisolone
Drug: Cytoxan — Alkylating agent, 100mg, 200 mg, and 500mg vials, and 1 and 2 gram vials, via intravenous (into the vein) infusion per institutional standard of care.
  Other Names: Cyclophosphamide; Cyclophosphamide-OE
Drug: Carmustine — Alkylating agent, 100 mg single dose vials, via intravenous (into the vein) infusion per institutional standard of care.
  Other Names: BiCNU
  Arms: Tazemetostat + CHOP Therapy + Transplant Elected
Drug: Etoposide — Topoisomerase II inhibitor, 100mg single dose vial, via intravenous (into the vein) infusion per institutional standard of care.
  Other Names: Etopophos
  Arms: Tazemetostat + CHOP Therapy + Transplant Elected
Drug: Cytarabine — Antineoplastic, 20mg single dose vial, via intravenous, intrathecal, or subcutaneous injection per institutional standard of care
  Arms: Tazemetostat + CHOP Therapy + Transplant Elected
Drug: Melphalan — Alkylating agent, 90 mg multi-dose vial, via parenteral infusion per institutional standard of care.
  Arms: Tazemetostat + CHOP Therapy + Transplant Elected

SUMMARY:
This research is being done to evaluate tazemetostat in combination with CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone) chemotherapy as a possible treatment for peripheral T-Cell Lymphoma (PTCL).

The name of the study drugs involved in this study are:

* Tazemetostat (a type of inhibitor for Enhancer of Zeste Homolog 2 (EZH2))
* Standard of care CHOP therapy:

  * Cyclophosphamide (a type of alkylating agent)
  * Doxorubicin (a type of anthracycline antibiotic)
  * Vincristine (a type of vinca alkaloid)
  * Prednisone (a type of corticosteroid)
* Standard of care BEAM conditioning regimen for autologous stem cell transplant:

  * Carmustine (a type of alkylating agent)
  * Etoposide (a type of Topoisomerase II inhibitor)
  * Cytarabine (a type of antineoplastic)
  * Melphalan (a type of alkylating agent)

DETAILED DESCRIPTION:
This is a phase 2 open-label study of Tazemetostat plus CHOP chemotherapy to find out if the addition of Tazemetostat is more beneficial than the usual approach for PTCL, which is CHOP or CHOEP (CHOP with Etoposide) with a potential standard-of-care autologous stem cell transplant. Tazemetostat works to slow down and decrease specific proteins that may be overactive in PTCL.

The U.S. Food and Drug Administration (FDA) has not approved tazemetostat for Peripheral T-Cell Lymphoma but it has been approved for other uses cancers including a different type of lymphoma called Follicular Lymphoma.

The FDA has approved CHOP as a treatment option for PTCL.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, electrocardiograms (ECGs), echocardiograms (Echos), Positron Emission (PET) scans, Computerized Tomography (CT) scans, tumor biopsies, and bone marrow biopsies and aspirations.

It is expected that about 24 people will take part in this research study.

Ipsen is supporting this research study by providing the study drug, tazemetostat and funding.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed peripheral T cell lymphoma of one of the following subtypes: PTCL-NOS, Follicular helper T-cell lymphoma (ICC 2022) or Nodal T-follicular helper (TFH) cell lymphoma by (WHO 2022) which includes follicular helper T-cell lymphoma, AITL and follicular helper T cell lymphoma, follicular type, EATL, MEITL. All pathology will be reviewed at BWH. BWH review is not required prior to enrollment and patients may be enrolled based upon local pathology analysis. Ten blank slides will be required from outside tumor biopsy for correlative studies.
* No prior treatment for T NHL with the exception of one cycle of CHOP or CHOEP or 7 days of corticosteroids at a dose of up to prednisone 60 mg or equivalent for palliation of disease related symptoms so long as the corticosteroids are discontinued prior to tazemetostat prephase or cycle 1 of treatment if not receiving the prephase.
* At least one bi-dimensionally measurable lesion, defined as >1.5 cm in its longest dimension as measured by CT.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/mcL (750 mcl if bone marrow involvement with lymphoma)
  * platelets ≥75,000/mcL (25,000 if bone marrow involvement with lymphoma)
  * total bilirubin ≤ institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * creatinine ≤ 1.5 x institutional ULN OR
  * glomerular filtration rate (GFR) ≥60 mL/min/1.73 m2
* Because the effects of tazemetostat on human immunodeficiency virus (HIV)-infected participants and anti-retroviral therapy is unknown, patients with known HIV infection are not eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment, are not eligible.
* Left ventricular ejection fraction of > 50% as assessed by echocardiography or multi-gate acquisition (MUGA) scan.
* The effects of tazemetostat on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. For women of childbearing potential, a negative serum pregnancy test result within 7 days prior to commencement of dosing. Women who are considered not to be of childbearing potential are not required to have a pregnancy test.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of tazemetostat administration.Women should use effective contraceptive methods beginning ≥28 days prior to initiating, during tazemetostat treatment, and for at least 6 months after the final dose of tazemetostat
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy for T cell lymphoma prior to entering the study (except 1 cycle of CHOP/CHOEP as noted above). Prior radiotherapy may be allowed after discussion with the sponsor-investigator so long as the area radiated was not the only measurable site of disease.
* Participants who are receiving any other investigational agents.
* Patients with known central nervous system involvement with lymphoma
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tazemetostat or other agents used in study.
* Prior organ transplantation.
* Current motor or peripheral neuropathy with grade >1.
* History of other malignancy that could affect compliance with the protocol or interpretation of results. Exceptions include:

  * Patients with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix at any time prior to the study are eligible.
  * Patients with any malignancy appropriately treated with curative intent and the malignancy has been in remission without treatment for > 2 years prior to enrollment are eligible.
  * Patients with low-grade, early-stage prostate cancer (Gleason score 6, Stage 1 or 2) with no requirement for therapy at any time prior to study are eligible.
* Uncontrolled intercurrent illness.
* Pregnant women and women intending to become pregnant are excluded from this study because chemotherapeutic agents used in this study have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with tazemetostat, breastfeeding should be discontinued if the mother is treated with tazemetostat.
* Evidence of significant, uncontrolled, concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina)
* Recent major surgery (within 4 weeks prior to the start of Cycle 1), other than for diagnosis
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or significant infections within 2 weeks before the start of Cycle 1.
* Inability to swallow pills.
* Because no dosing or adverse event data are currently available on the use of tazemetostat in combination with CHOP in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | Up to 18 weeks
  CRR rate was defined as the proportion of participants who achieved CR during the first six cycles of treatment.

SECONDARY OUTCOMES:
Median Overall Survival (OS) | Up to 5.5 years
  OS based on Kaplan-Meier methodology is defined as the time from registration to death due to any cause, or censored at date last known alive.
Median Progression Free Survival (PFS) | Up to 1.5 years
  PFS based on the Kaplan-Meier method is defined as the time from first study treatment to the first occurrence of disease progression or relapse as assessed or death from any cause, whichever occurs earlier. Confirmation of progression by biopsy is preferred.
Duration of Response (DOR) | Up to 1.5 years
  The duration of overall response is defined as the time from first documentation of PR to CR until first documentation of progression or relapse by clinical or radiology parameters. Confirmation of progression by biopsy is preferred. Participants without events reported are censored at the last disease evaluation.
Grade 3-5 Treatment-Related Toxicity Rate | Up to 3.5 years
  The percentage of participants who experienced a maximum grade 3-5 treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.
Transplant Rate | Up to 1.5 years
  Transplant rate defined as the proportion of participants who are deemed transplant eligible and nominated by the treating investigator before initiation of protocol therapy to undergo consolidation transplant, who receive at least one dose of protocol-based therapy, and who then successfully proceed to transplant.
Mobilization Success Rate | Up to 1.5 years
  Mobilization success rate is defined as the proportion of participants nominated by the treating investigator before initiation of protocol therapy to undergo consolidation transplant, in whom stem cell mobilization is attempted and who mobilize a sufficient number of stem cells to proceed to stem cell transplant irrespective of actually proceeding to transplant. Mobilization success will be determined by institutional standards for absolute number of CD34+ cells necessary for transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu